CLINICAL TRIAL: NCT02018822
Title: Clinical Evaluation of an Experimental Urethane Dimethacrylate Resin Based Composite
Brief Title: Evaluate the Effectiveness of an Experimental Urethane Dimethacrylate Resin Based Dental Composite Material
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Hans Malmstrom, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 765-552
Record Dates: First submitted 2013-12-17; First posted 2013-12-23 (Estimated); Results first posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-07

CONDITIONS: Dental Caries; Restorative Material
Keywords: restorative material
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Participants (Experimental): Participants who needed at least two tooth restorations
  Interventions: Device: urethane dimethacrylate; Device: TPH3; Device: Esthet-X HD

INTERVENTIONS:
Device: urethane dimethacrylate — Experimental urethane dimethacrylate resin based composite resin for teeth used with prime and Bond Elect bonding agent
Device: TPH3 — light-cured resin composite for teeth
Device: Esthet-X HD — light cured resin composite for teeth made by Dentsply Caulk

SUMMARY:
This double blind randomized controlled prospective clinical trial will compare the clinical success of two tooth colored resin composite dental filling materials - TPH3 (Dentsply Caulk) and an experimental urethane dimethacrylate resin based composite resin (Dentsply Caulk) for wear resistance, staining and marginal seal using modified Ryge criteria to evaluate the posterior restorations for 24 months in duration

DETAILED DESCRIPTION:
The purposes of this clinical trial is to evaluate two composite resins used to restore Class I and Class II cavities in teeth of adults. The clinical study will evaluate the resin composite restorations placed in Class I and Class II cavity preparations for anatomic form, color match, marginal integrity, marginal discoloration, proximal contact, polishability, caries, sensitivity, gingival index, staining,wear, and thermal response for 24 months..

ELIGIBILITY:
Inclusion Criteria:• must have given written consent to participate in the trial

* must be in need of at least two restorations in natural tooth
* replacement restorations with or without caries are acceptable
* must be available for the required post-operative follow-up visits
* restorations to be in bicuspids, 1st or 2nd molars
* restorations to be in contact with opposing natural or crowned teeth
* class II restorations must have at least one proximal contact
* restorations must have a buccal to lingual/palatal width equal to or greater than 1/3 the distance from buccal to lingual/palatal cusp tips
* 75% of the restorations must be Class II
* all restorations must have at least one occlusal contact in habitual closure

Exclusion Criteria:

* have severe medical complications (organ transplants, long term antibiotic or steroid treatment, cancer or immunocompromised) or disabilities who may not be able to tolerate the time required to complete the restorations or to provide adequate oral hygiene
* have xerostomia either by taking medications known to produce xerostomia or those with radiation induced or Sjogren's syndrome patients
* have chronic periodontitis, rampant caries or poor oral hygiene which may require extraction of the teeth to be restored
* have a history of chronic bruxism and those unavailable for long term recall
* can not tolerate the rubber dam required for tooth isolation during preparation and restoration.
* do not meet all inclusion criteria
* present with any systemic or local disorders that contra-indicate the dental procedures included in this study
* have an unstable occlusion
* have severe bruxing or clenching or need of TMJ related therapy
* have teeth with periapical pathology or expected pulp exposures
* have teeth that are non-vital or that exhibit signs of pulpal pathology
* Pregnancy
* Known sensitivity to methacrylates and/or acrylates

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-06; Primary Completion 2017-06-29 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Eastman Institute for Oral Health, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 participants received both TPH3 and UDMA in a split-face design, with the most anterior or right tooth randomized to one intervention and the most posterior or left tooth randomized to the second intervention. An additional 35 participants were included for treatment with Esthet-X and could receive the intervention on more than one tooth.
Units Other Than Participants: teeth
Groups:
- UDMA: Participants who needed at least two tooth restorations
  urethane dimethacrylate: Experimental urethane dimethacrylate resin based composite resin for teeth used with prime and Bond Elect bonding agent
  TPH3: light-cured resin composite for teeth
  Esthet-X HD: light cured resin composite for teeth made by Dentsply Caulk
- TPH3: Participants who needed at least two tooth restorations
  TPH3: light-cured resin composite for teeth
- Esthet-X: Participants who needed at least two tooth restorations
Period: Overall Study
Arm/Group | UDMA | TPH3 | Esthet-X
Started | 50; 50 teeth | 50; 50 teeth | 35; 50 teeth
Completed (Completed 24 months) | 44; 44 teeth | 42; 42 teeth | 29; 41 teeth
Not Completed | 6; 6 teeth | 8; 8 teeth | 6; 9 teeth
Not completed — filling replaced by crown | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 1
Not completed — Lost to Follow-up | 6 | 6 | 5

BASELINE CHARACTERISTICS:
Population: 50 participants were enrolled. Each received the UDMA and TPH3 interventions. 35 were enrolled to recieve the Esthet-X intervention.
Groups:
- UDMA and TPHs; Esthet-X HD: Participants who needed at least two tooth restorations
- Total: Total of all reporting groups
Arm/Group | UDMA and TPHs | Esthet-X HD | Total
Number analyzed (Participants) | 50 | 35 | 85
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 35 | 85
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 23 | 59
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 3 | 12
  Not Hispanic or Latino | 41 | 31 | 72
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 3 | 9
  White | 42 | 27 | 69
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 35 | 85

OUTCOME MEASURES:

1. Primary Outcome: Percent of Teeth With Anatomic Form Graded as A or B.
Description: Anatomic form was graded as:
  A=The restoration is continuous with existing form. B=The restoration is discontinuous with existing anatomic form, but the existing material is not sufficient to expose dentine.
Time Frame: 24 months
Population: Participants with available data at 24 months. Two participants who received both the UDMA and TPH3 interventions were unevaluable for the TPH3 intervention at this time point.
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Groups:
- Teeth That Received UDMA: Experimental urethane dimethacylate resin based composite for teeth used with prime and Bond Elect bonding agent
- Teeth That Received TPH3: light-cured resin composite for teeth
- Teeth That Received Esthet-X-HD: light cured resin composite for teeth made by Dentsply Caulk
Arm/Group | Teeth That Received UDMA | Teeth That Received TPH3 | Teeth That Received Esthet-X-HD
Number analyzed (Participants) | 44 | 42 | 29
Number analyzed (teeth) | 44 | 42 | 41
teeth
  A | 42 | 37 | 40
  B | 2 | 5 | 1
Statistical Analysis 1: Comparison: Teeth That Received UDMA vs Teeth That Received TPH3 vs Teeth That Received Esthet-X-HD; Test type: Non-Inferiority — Assuming that the success rate of the control composite resin is 95% based on clinical data, for a non-inferiority test with a non-inferiority margin of 15%, a sample size of 27 is required in each group to allow 80% power at an alpha level of 0.05. We aimed to have 30 subjects/teeth remaining in each group after attrition at the end of the study; p = 0.2552, Chi-squared

2. Primary Outcome: Percent of Teeth Scored as A or B for Color Match
Description: A=The restoration appears to match the shade and translucency of adjacent tooth structure.
  B=The restoration does not match the shade and translucency of adjacent tooth structure, but the mismatch is within the normal range of tooth shades and translucency.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Groups:
- UDMA: Experimental urethane dimethacylate resin based composite for teeth used with prime and Bond Elect bonding agent
- Participants That Completed Esthet-X Intervention: light cured resin composite for teeth made by Dentsply Caulk
Arm/Group | UDMA | TPH3 | Participants That Completed Esthet-X Intervention
Number analyzed (Participants) | 44 | 42 | 29
Number analyzed (teeth) | 44 | 42 | 41
teeth
  A | 41 | 40 | 40
  B | 3 | 2 | 1
Statistical Analysis 1: Comparison: UDMA vs TPH3 vs Participants That Completed Esthet-X Intervention; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.2235, Chi-squared

3. Primary Outcome: Percent of Teeth With Marginal Integrity Graded A, B1 and B2
Description: A= No visible evidence of a crevice along the margin into which the explorer will penetrate B1= Explorer clicks on the margin B2= Visible evidence of a crevice
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Teeth That Received UDMA | Teeth That Received TPH3 | Teeth That Received Esthet-X-HD
Number analyzed (Participants) | 44 | 42 | 29
Number analyzed (teeth) | 44 | 42 | 41
teeth
  A | 39 | 36 | 39
  B1 | 2 | 4 | 1
  B2 | 3 | 2 | 1
Statistical Analysis 1: Comparison: Teeth That Received UDMA vs Teeth That Received TPH3 vs Teeth That Received Esthet-X-HD; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3891, Chi-squared

4. Primary Outcome: Percent of Teeth With Marginal Discoloration of A or B
Description: A= There is no visual evidence of marginal discoloration different from the color of the restorative material and from the color the adjacent tooth structure.
  B= There is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration, but the discoloration has not penetrated along the restoration in a pulpal direction.
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Teeth That Received UDMA | Teeth That Received TPH3 | Teeth That Received Esthet-X-HD
Number analyzed (Participants) | 44 | 42 | 29
Number analyzed (teeth) | 44 | 42 | 41
teeth
  A | 39 | 40 | 39
  B | 5 | 2 | 2
Statistical Analysis 1: Comparison: Teeth That Received UDMA vs Teeth That Received TPH3 vs Teeth That Received Esthet-X-HD; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3883, Chi-squared

5. Primary Outcome: Percent of Teeth With Proximal Contact
Description: A= Tight proximal contacts evaluated with dental floss. B= Proximal contacts are weak but present. C= No proximal contacts but not visibly open. NA= Class I restorations
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Teeth That Received UDMA | Teeth That Received TPH3 | Teeth That Received Esthet-X-HD
Number analyzed (Participants) | 44 | 42 | 29
Number analyzed (teeth) | 44 | 42 | 41
teeth
  A | 32 | 28 | 29
  B | 4 | 4 | 2
  C | 1 | 1 | 0
  NA | 7 | 9 | 10
Statistical Analysis 1: Comparison: Teeth That Received UDMA vs Teeth That Received TPH3 vs Teeth That Received Esthet-X-HD; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.3883, Chi-squared

6. Primary Outcome: Percent of Teeth With Polish-ability of A, B1 or B2
Description: A= Smooth & highly shiny, similar to enamel B1= Smooth & satin, highly reflective B2= Smooth & shiny but not highly reflective
Time Frame: 24 months
Population: as for outcome 1
Measure: Count of Units; unit: teeth
Units Other Than Participants: teeth
Arm/Group | Teeth That Received UDMA | Teeth That Received TPH3 | Teeth That Received Esthet-X-HD
Number analyzed (Participants) | 44 | 42 | 29
Number analyzed (teeth) | 44 | 42 | 41
teeth
  A | 41 | 40 | 40
  B1 | 2 | 1 | 1
  B2 | 1 | 1 | 0
Statistical Analysis 1: Comparison: Teeth That Received UDMA vs Teeth That Received TPH3 vs Teeth That Received Esthet-X-HD; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.2707, Chi-squared

ADVERSE EVENTS:
Time Frame: 24 months
Groups:
- UDMA: Experimental urethane dimethacrylate resin based composite resin for teeth used with prime an Bond Elect bonding agent
Arm/Group | UDMA | TPH3 | Esthet-X HD
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50 | 0/35
Other Adverse Events (participants affected / at risk) | 0/50 | 2/50 | 1/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UDMA (N=50) | TPH3 (N=50) | Esthet-X HD (N=35)
No response on tooth vitality test (General disorders) | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT02018822/Prot_SAP_000.pdf